CLINICAL TRIAL: NCT03234088
Title: Home Based Health Monitoring for Congestive Heart Failure Pilot
Brief Title: Congestive Heart Failure Pilot Study Utilizing Wireless Home Scale and Daily Symptom Monitoring
Acronym: CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC2AG036592 (NIH)
Record Dates: First submitted 2011-01-21; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Heart Failure; Home telemonitoring; Telehealth; HF Disease Management; Heart failure remote self management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home HF monitoring (Other): Digital scale readings are transmitted wirelessly to the handheld device. Patients will remotely log on to a secure server to answer daily symptom questions. Patients will complete surveys after voluntarily completing the informed consent process and at study closeout.
  Interventions: Behavioral: Daily weight measured by digital scale and symptom reporting

INTERVENTIONS:
Behavioral: Daily weight measured by digital scale and symptom reporting — All subjects will be provided the intervention.
  Other Names: MedApps Healthcom wireless digital scale is being utilized

SUMMARY:
As the population ages and medicine advances, there has been a significant shift to the management of chronic diseases. Most chronic diseases are managed using evidence based consensus guidelines but clinician and patient compliance with these guidelines is sub-optimal. In addition, due to the nature of chronic diseases, patients need to make long-term lifestyle changes in order to effectively control their disease in order to minimize complications, disability and cost. It is these two factors, consistent implementation of evidence-based guidelines and supporting patients in a way that encourages self-management and lifestyle change, that disease management attempts to impact. There are areas of design, implementation, testing and final-result-reporting to the patient and clinician that require collaboration among information technology (IT) and software design engineers and clinicians to achieve several goals:

1. Ensure patient safety.
2. Protect the security and integrity of clinical data.
3. Provide patient specific education to promote self-management.
4. Provide actionable data to clinicians in order to improve clinical care and minimize the risk of adverse events.
5. Provide both patient and clinician satisfaction with the system of care.

In order to achieve these goals, testing and development of home technology under a controlled clinical trial is critical.

DETAILED DESCRIPTION:
This study will consist of: Specific Aim 1, Perform a pilot study to evaluate the initial performance of the wireless scale and symptom monitoring system on a select number of presumed normal volunteers (five). The purpose of this will be to determine design and process changes prior to the use of the device in subjects with chronic heart failure (HF). The investigators will have each normal volunteer (all part of the key research team) perform scenarios to test the performance of the system. Specific Aim 2 will incorporate changes into the prototype system adapting both the technology as well as the clinical workflows surrounding its use based on the information collected in Specific Aim 1. Specific Aim 3 will evaluate the revised system enrolling 40 volunteer subjects that have provided written voluntary consent with the documented primary diagnosis of HF (systolic or diastolic) to participate in the intervention over a 4-month period with the primary outcome measure being reduction in HF related ER visit or hospitalization.

The objective of this study is to pilot test and refine a new home-based telemedicine health monitoring system that provides wireless, low cost measurement of body weight as well as self-reported responses, including symptoms and medication compliance for the purpose of managing chronic heart failure (HF) within the home. This pilot will test the functionality of the research infrastructure first on 5 healthy volunteers and then on 40 patients with heart failure over 4 months, testing the receipt of accurate input from the wireless scale and then assessing the effectiveness of the scale intervention in reducing ER visits and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of heart failure (either systolic or diastolic) NYHA class II, III and IV
* Physical and cognitive ability to use the device
* Cellular phone or other portable device with "text" communication capability or daily access to the internet using a computer or laptop

Exclusion Criteria:

* Subject with life expectancy less than 6 months from any cause, or enrolled in hospice care.
* Subject not competent or unwilling to give voluntary informed consent.
* Subject currently participating in another home telemedicine intervention trial
* Subjects with a left ventricular assist device or who have had a cardiac transplant
* Dialysis upon screening or creatinine >2.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Usage of home-health monitoring devices for weight | Baseline through study completion, an average of four months
  Monitoring daily weights and heart failure symptoms

SECONDARY OUTCOMES:
Patient and Provider Questionnaires on usability and functionality of the study's online web portal (Way to Health) | Baseline through study completion, an average of four months
Patient and Provider Questionnaires on usability and functionality of the study's wifi-enabled home health monitoring devices | Baseline through study completion, an average of four months

CONTACTS AND LOCATIONS:
Overall Officials: Lee R Goldberg, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Caveat emptor: the need for evidence, regulation, and certification of home telehealth systems for the management of chronic conditions. — http://www.ncbi.nlm.nih.gov/pubmed/18539982?dopt=AbstractPlus
- See also: Randomized trial of a daily electronic home monitoring system in patients with advanced heart failure: the Weight Monitoring in Heart Failure (WHARF) trial. — http://www.ncbi.nlm.nih.gov/pubmed/14564327
- See also: Validation of prognostic models among patients with advanced heart failure. — http://www.ncbi.nlm.nih.gov/pubmed/16911909
- See also: Electronic and telemedicine techniques to manage heart failure. — http://www.ncbi.nlm.nih.gov/pubmed/16004864
- See also: Baseline differences in the HF-ACTION trial by sex. — http://www.ncbi.nlm.nih.gov/pubmed/19782784